CLINICAL TRIAL: NCT03404635
Title: Monotherapy Anticoagulation To Expedite Home Treatment of Venous
Brief Title: Monotherapy Anticoagulation To Expedite Home Treatment of Venous Thromboembolism
Acronym: MATHVTE
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Pfizer (Industry); Janssen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Jeffrey Kline, Professor of Emergency Medicine, Indiana University
Other Study IDs: CV185-562
Record Dates: First submitted 2017-12-19; First posted 2018-01-19 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Apixaban for VTE
  Interventions: Drug: Apixaban
- Rivaroxaban for VTE
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Apixaban — Apixaban as standard of care for VTE
  Groups: Apixaban for VTE
Drug: Rivaroxaban — Rivaroxaban as standard of care for VTE
  Groups: Rivaroxaban for VTE

SUMMARY:
Prospective, multicenter observational study, of the effectiveness of a standard of care protocol implemented to enhance home treatment of VTE. Study population will be selected as part of usual care as eligible for home treatment. Study personnel will travel to participating institutions to qualify the sites, deliver a Powerpoint® lecture to introduce the protocol, meet and train site principal investigators, emergency physicians and research personnel on the implementation of the protocol as part of usual clinical care, and data collection methods for a quality assurance registry with plans to use the data collected in this registry in future publications. Follow-up will be 30 days using medical records and/or telephone interview to assess for primary outcomes of bleeding or VTE recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be low risk, as defined by either A or B below:

   A. The modified Hestia criteria:
   * Systolic blood pressure > 100 mm Hg
   * No thrombolysis needed
   * No active bleeding
   * SaO2 >94% while breathing room air
   * Not already anticoagulated
   * No more than two doses of IV narcotics in the emergency department
   * Other medical or social reasons to admit
   * Creatinine clearance >30mL/min
   * Not pregnant, severe liver disease or heparin induced thrombocytopenia OR

   B. The physician opinion that a patients' overall social and medical situation is favorable for home treatment and the patient has a zero score on the simplified pulmonary embolism severity index (sPESI).

   All of the following must true:
   * Age < 81 years
   * No history of cancer
   * No history of heart failure or chronic lung disease
   * Pulse < 110 beats/min
   * SBP > 99 mm Hg
   * O2 sat >89%%

   We have chosen either criteria because both have been found equal in terms of safety for outpatient treatment of PE.6,22 Hestia includes implicit questions that most emergency physicians would use as criteria for discharge (e.g., overall medical status and social situation), whereas sPESI does not. For that reason, we have added the additional gestalt assessment question about physician discretion.
2. Patients must be discharged in <24 hours after triage in an ED visit with diagnosis of VTE using objective criteria in the emergency department.

Exclusion Criteria:

* VTE diagnosis while taking anticoagulants with evidence of compliance (e.g., physician opinion that patient is taking a Eliquis®, Xarelto® or Pradaxa®, low molecular weight heparin injections or warfarin as prescribed for any condition)
* Sensitivity or contraindication to use of apixaban
* Troponin assay value, drawn as part of usual care and found to be positive, using local standards
* High risk for hemorrhage defined by a score>1.5 using the method of Ruiz Gimenez.3 (Note that several criteria are already excluded by Hestia):

Recent major bleeding, 2 points Creatinine levels >1.2 mg/dl, 1.5 points Anemia, 1.5 points Cancer, 1 point Clinically overt PE, 1 point Age >75 years, 1 point

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patients with new or recurrent VTE deemed low-risk by modified Hestia or clinician discretion and sPESI (-).
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Number of re-hospitalization visits for VTE recurrence or bleeding | 30 days
  Re-hospitalization for > 24 hours due to VTE recurrence or bleeding

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Eskenazi Health System, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kline JA, Adler DH, Alanis N, Bledsoe JR, Courtney DM, d'Etienne JP, Diercks DB, Garrett JS, Jones AE, Mackenzie DC, Madsen T, Matuskowitz AJ, Mumma BE, Nordenholz KE, Pagenhardt J, Runyon MS, Stubblefield WB, Willoughby CB. Monotherapy Anticoagulation to Expedite Home Treatment of Patients Diagnosed With Venous Thromboembolism in the Emergency Department: A Pragmatic Effectiveness Trial. Circ Cardiovasc Qual Outcomes. 2021 Jul;14(7):e007600. doi: 10.1161/CIRCOUTCOMES.120.007600. Epub 2021 Jun 21. PMID 34148351